CLINICAL TRIAL: NCT01876693
Title: A Prospective Study of Prophylactic Gastrostomy in Head and Neck Cancer Patients Undergoing Chemoradiotherapy in Medical Practice
Brief Title: A Prospective Study of Prophylactic Gastrostomy in Head and Neck Cancer Patients Undergoing Chemoradiotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual in experiment arm
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, suthinee ithimakin, Assistant professor, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: si041/2013
Record Dates: First submitted 2013-05-21; First posted 2013-06-12 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): nutrition counselling with nasogastric tube insertion in the cases of weight loss more than 10% or severe mucositis developed during chemoradiotherapy
- prophylactic percutaneous gastrostomy (Experimental): prophylactic percutaneous gastrostomy with nutrition counselling
  Interventions: Procedure: prophylactic percutaneous gastrostomy

INTERVENTIONS:
Procedure: prophylactic percutaneous gastrostomy — prophylactic percutaneous gastrostomy with nutrition counselling
  Arms: prophylactic percutaneous gastrostomy

SUMMARY:
The purpose of the study is to determine whether prophylactic gastrostomy leads to less treatment interruption and provide better quality of life in head and neck cancer patients receiving chemoradiotherapy.

DETAILED DESCRIPTION:
Nutritional status is one of the essential factor to determine outcome of chemoradiotherapy in head and neck cancer patients. Almost all these patients develop mucositis during the treatment, which usually leads to treatment interruptions and affects the efficacy of the treatment. Prophylactic gastrostomy has been accepted for these patients with improvement of quality of life. However, there is no prospective study confirming superiority of such treatment.

The investigators enrolled head and neck cancer patients who had the plan of chemoradiotherapy. The patients will be informed about both treatment arms and will decide the arm that they preferred. The treatment interruptions, body weight and nutritional status will be assessed every 2 weeks during treatment period.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed of head and neck cancer
* plan to have chemoradiotherapy session
* Performance status of 0-2

Exclusion Criteria:

* contraindications for percutaneous gastrostomy, eg coagulopathy, obstructed tumor
* Body mass index less than 16 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
treatment interruption due to toxicity | during period of chemoradiatherapy, an expected average of 6 weeks

SECONDARY OUTCOMES:
quality of life | during period of chemoradiation, an expected avearage of 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suthinee Ithimakin, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Division of medical oncology, department of medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pramyothin P, Manyanont S, Trakarnsanga A, Petsuksiri J, Ithimakin S. A prospective study comparing prophylactic gastrostomy to nutritional counselling with a therapeutic feeding tube if required in head and neck cancer patients undergoing chemoradiotherapy in Thai real-world practice. J Hum Nutr Diet. 2016 Dec;29(6):768-776. doi: 10.1111/jhn.12377. Epub 2016 Mar 29. PMID 27028666